CLINICAL TRIAL: NCT00681707
Title: A Retrospective, Multi Centre, Non-Interventional, Observational Study to Investigate Treatment Pattern of Blood Pressure in the Post Stroke Patients With Hypertension.
Brief Title: Retrospective Treatment Pattern Survey for the Patients With Hypertension and Stroke
Acronym: SAPPHIRE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Joonwoo Bahn, AstraZeneca
Other Study IDs: NIS-CKR-DUM-2008/1
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
Keywords: Hypertension; Post stroke; JNC7; 2007 ESH-ESC guidelines; survey
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Hypertension patients recovering from stroke

SUMMARY:
This study will address the treatment rate and control rate of hypertension, treatment pattern and factors that affect BP control by examining retrospective medical records of hypertension patients recovering from stroke, among outpatients coming to the Neurology Department in 10 university hospitals nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Patients had been hospitalized as a acute stroke in 2006
* Patient with history of stroke receiving hypertension medication during at least 1 year.

Exclusion Criteria:

* Secondary hypertension patients
* Patients not receiving hypertension medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with history of stroke, receiving hypertension medication during at least 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-05; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Attainment rate to the target blood pressure | After collecting all Patient Record Form.

SECONDARY OUTCOMES:
Dropout rate will be estimated during the follow-up period after the hypertension treatment. Attainment to the target blood pressure will be investigated according to concomitant diseases. | After collecting all Patient Record Form.
Change in DBP/SBP value during the follow-up period will be addressed. Change in the DBP/SBP value will be investigated according to the risk factors and concurrent disease. | After collecting all Patient Record Form.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Woo Bahn, Study Director — Astrazenca Korea medical dept.
Locations (8):
- South Korea (8):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Sungnam, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Deagu
  - Research Site, Deajeon
  - Research Site, Kwangju
  - Research Site, Seoul